CLINICAL TRIAL: NCT05026892
Title: Identification of Factors Associated With the Occurrence of Severe Forms of COVID-19 Infection in Patients With Inflammatory Rheumatism or Autoimmune Diseases
Acronym: CovAID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: FAI²R (Auto-immune and auto-inflammatory rare diseases French network) (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP200714
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV2 Infection; Rare Diseases; Chronic Inflammatory Rheumatism; Autoimmune Diseases
Keywords: SARS-CoV2 Infection; Rare Diseases; Chronic Inflammatory Rheumatism; Autoimmune Diseases; auto-inflammatory diseases
MeSH Terms: conditions — COVID-19; Rare Diseases; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- moderate to severe: patients with known inflammatory rheumatism, auto-immune or auto-inflammatory diseases (as define in the inclusion criteria) with moderate to severe or severe form of covid-19
  Interventions: Other: no intervention
- begining to moderate: Patients with known inflammatory rheumatism, auto-immune or auto-inflammatory diseases (as define in the inclusion criteria) with begnin to moderate or moderate form of covid-19
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, only collection of data

SUMMARY:
Factors associated with severe forms of COVID-19 infection in patients with inflammatory rheumatic diseases (IRD) or Autoimmune Diseases (AID) are unknown. This unprecedented situation leads to empirical and potentially erroneous advice and recommendations for care. Identifying factors associated with severity, in the context of this pandemic, which is expected to last many months, and possibly years, is crucial for future patients. The objective of this work is to identify the factors associated with the occurrence of severe forms of COVID-19 infection in patients with IRD or AID, by combining analysis of 2 large databases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known chronic inflammatory rheumatism, auto-immune or auto-inflammatory diseases (Rheumatoid arthritis, Spondyloarthritis, Psoriatic arthritis Lupus, Sjögren's syndrome, Inflammatory Myositis, Systemic Vasculitis, Sarcoidosis, Scleroderma, PPR/Horton's, other ...)
* At least 18 years old
* SARS-Cov-2 infection (COVID-19) by biological data (serological or positive Cov-2 PCR) or CT scan images or clinical observations consistent with covid-19 between January 2020 and September 2020
* data available in the APHP health data center (EDS) or in the french RMD Covid19 cohort

Exclusion Criteria:

* patients opposed to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known chronic inflammatory rheumatism, auto-immune or auto-inflammatory diseases (Rheumatoid arthritis, Spondyloarthritis, Psoriatic arthritis Lupus, Sjögren's syndrome, Inflammatory Myositis, Systemic Vasculitis, Sarcoidosis, Scleroderma, PPR/Horton's, other ...) with confirmed SARS-Cov-2 infection (COVID-19) whose data are available in the APHP health data center (EDS) or in the french RMD Covid19 cohort
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
risk factors associated with severity | during covid infection
  Between begining to moderate and moderate to severe group: Severe form is defined by be defined by hospitalization in intensive care unit and/or death. Demographic, Comorbidities (and their treatments), underlying IRD and AID and treatments for IRD or AID will be analysed.

SECONDARY OUTCOMES:
risk factors associated with severe form | during covid infection
  in moderate to severe group: Moderate to severe form is defined by be defined by hospitalization for COVID infection. Demographic, Comorbidities (and their treatments), underlying IRD and AID and treatments for IRD or AID will be analysed. Pooled analysed and Analyses by IRD/AID subset will be performed, since prognosis might differ in the different diseases : IRD (including rheumatoid arthritis and spondyloarthritis), other AID, and systemic vaculitis)
risk factors associated with severe form | during covid infection
  in severe group only: Severe form is defined by be defined by hospitalization in intensive care unit and/or death. Demographic, Comorbidities (and their treatments), underlying IRD and AID and treatments for IRD or AID will be analysed. Analyses by IRD/AID subset will be performed, since prognosis might differ in the different diseases : IRD (including rheumatoid arthritis and spondyloarthritis), other AID, and systemic vaculitis)
risk factors associated with death | during covid infection
  Death during COVID-19 infection. Demographic, Comorbidities (and their treatments), underlying IRD and AID and treatments for IRD or AID will be analysed. Pooled analysed and Analyses by IRD/AID subset will be performed, since prognosis might differ in the different diseases : IRD (including rheumatoid arthritis and spondyloarthritis), other AID, and systemic vaculitis)

CONTACTS AND LOCATIONS:
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France